CLINICAL TRIAL: NCT06593561
Title: Turkish Version of Breast Edema Questionnare: Validity and Reliability Study
Status: Completed | Type: Observational
Sponsor: Aysima Barlak (Other)
Responsible Party: Sponsor-Investigator, Aysima Barlak, PT, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: GO22/879
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-02

CONDITIONS: Breast Edema
Keywords: radiotherapy; breast cancer; lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Breast Edema Questionnare — The Breast Edema Questionnaire, developed to evaluate breast edema in women undergoing breast cancer surgery, will be applied.

SUMMARY:
This study was planned to investigate the complaint of breast edema after breast conserving surgery and radiotherapy, which are considered as the main treatment modalities for breast cancer. The incidence of breast edema after these treatments ranges from 0% to 90.4%. In contrast to arm lymphedema, which has been described in detail in the literature, only a few studies have investigated breast edema. There is no survey study that comprehensively examines the presence of lymphedema and its clinical features (duration, severity, location). Studies to assess breast edema after breast cancer treatment have revealed the need for a condition-specific scale. Therefore, the "Breast Edema Questionnaire" was developed to assess breast edema in women who have undergone breast cancer surgery. The original language of this questionnaire is German and its reliability and validity has not been studied in another language. In this study, the validity and reliability of this questionnaire, which specifically assesses breast edema, will be tested in Turkish women.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of breast cancer who have undergone breast-conserving surgery
* individuals who have signed the Informed Consent form

Exclusion Criteria:

* illiterate individuals

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female individuals diagnosed with breast cancer, undergoing breast conserving surgery, literate, and signed the informed consent form will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Breast Edema Questionnare | one week
  Unlike arm lymphedema, which is described in detail in the literature, there are only a few studies investigating breast lymphedema after breast cancer treatment. Breast ultrasound (US) is considered to be a more reliable and quantitative measure of breast edema. However, there is no survey study that comprehensively examines these outcome measures according to the presence and clinical features of lymphedema (duration, severity, location of lymphedema). In studies conducted to evaluate breast edema after breast cancer treatment, the necessity of a situation-specific scale has emerged. For this reason, the "Breast Edema Questionnaire" was developed to evaluate breast edema in women undergoing breast cancer surgery.

SECONDARY OUTCOMES:
Ultrasound | baseline
  Ultrasonography is routinely used in the evaluation of skin and soft tissue complaints.Generally, ultrasound is used to evaluate abscesses, cellulitis and foreign bodies in the skin and soft tissue. The deterioration of the skin by bacterial invasion causes infection in the dermis and subcutaneous fat. These findings are due to subcutaneous edema accumulation. Ultrasound will be used to determine the localization, severity and amount of edema.
Moisture Meter Compact | baseline
  Fluid percentage will be evaluated using the Moisture Meter Compact instrument (Delphin technologies). The tissue dielectric constant (TDC) technique gives information about the emergence of lymphedema in the early stages and the change in the amount of water under the skin. The reflected wave contains information about the energy attraction, that is, the amount of water molecules in the skin. The resulting values are automatically converted to PWC values by the device software. The probe of the device showing the tissue dielectric constant will be placed on the skin. Tissue edema will be measured at different depths by making three different measurements. The reference point will be used.
Visual Analog Scale | baseline
  The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For example, for pain, I have no pain at one end and very severe pain at the other end and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy and Rehabilitation, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No